CLINICAL TRIAL: NCT00688740
Title: A Multicenter Phase III Randomized Trial Comparing Docetaxel in Combination With Doxorubicin and Cyclophosphamide (TAC) Versus 5-fluorouracil in Combination With Doxorubicin and Cyclophosphamide (FAC) as Adjuvant Treatment of Operable Breast Cancer Patients With Positive Axillary Lymph Nodes.
Brief Title: Docetaxel in Node Positive Adjuvant Breast Cancer
Acronym: TAX316
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Cancer International Research Group (CIRG) (Other)
Responsible Party: ICD Study Director, Sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC6041; XRP6976D-316; BCIRG001
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Results first posted 2011-02-14 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: Breast Cancer
Keywords: adjuvant treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Fluorouracil; Doxorubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAC (Docetaxel) (Experimental): docetaxel (75 mg/m^2) in combination with doxorubicin (50 mg/m^2) and cyclophosphamide (500 mg/m^2) on day 1 every 3 weeks for 6 cycles of treatment
  Interventions: Drug: Docetaxel; Drug: Doxorubicin; Drug: Cyclophosphamide
- FAC (5-fluorouracil) (Active Comparator): 5-fluorouracil (500 mg/m^2) in combination with doxorubicin (50 mg/m^2) and cyclophosphamide (500 mg/m^2) on day 1 every 3 weeks for 6 cycles of treatment
  Interventions: Drug: 5-fluorouracil; Drug: Doxorubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Docetaxel — intravenous
  Other Names: Taxotere®
  Arms: TAC (Docetaxel)
Drug: 5-fluorouracil — intravenous
  Other Names: 5-FU
  Arms: FAC (5-fluorouracil)
Drug: Doxorubicin — intravenous
Drug: Cyclophosphamide — intravenous

SUMMARY:
The purpose of this study was to compare disease-free survival after treatment with docetaxel in combination with doxorubicin and cyclophosphamide to 5-fluorouracil in combination with doxorubicin and cyclophosphamide in operable breast cancer patients with positive axillary lymph nodes.

DETAILED DESCRIPTION:
In addition to the 5-year analysis conducted in September 2003, two other analyses were planned when 590 and 700 Disease Free Survival events occurred. However, due to the lower than predicted DFS event rate, and in agreement with FDA and EMA, a time-based final analysis at 10 years was considered more appropriate than an event-based (700 Disease Free Survival events) analysis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven breast cancer (invasive adenocarcinoma with at least one axillary lymph node showing evidence of tumor among a minimum of six resected lymph nodes).
* Definitive surgical treatment must be either mastectomy, or breast conserving surgery with axillary lymph node dissection for operable breast cancer. Margins of resected specimen from definitive surgery must be histologically free of invasive adenocarcinoma and ductal carcinoma.

Exclusion criteria:

* Prior systemic anticancer therapy for breast cancer (immunotherapy, hormonotherapy, chemotherapy).
* Prior anthracycline therapy or taxoids (paclitaxel, docetaxel) for any malignancy.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1491 (Actual)
Dates: Start 1997-06; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ICD, Study Director — Sanofi
Locations (20):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Cairo, Egypt
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Berlin, Germany
- Sanofi-Aventis Administrative Office, Athens, Greece
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- sanofi-aventis Administrative office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Porto Salvo, Portugal
- Sanofi-Aventis Administrative Office, Bratislava, Slovakia
- Sanofi-Aventis Administrative Office, Midrand, South Africa
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-aventis adminsitrative office, Guildford Surrey, United Kingdom
- Sanofi-aventis administrative office, Montevideo, Uruguay

REFERENCES:
- [Result] Martin M, Pienkowski T, Mackey J, Pawlicki M, Guastalla JP, Weaver C, Tomiak E, Al-Tweigeri T, Chap L, Juhos E, Guevin R, Howell A, Fornander T, Hainsworth J, Coleman R, Vinholes J, Modiano M, Pinter T, Tang SC, Colwell B, Prady C, Provencher L, Walde D, Rodriguez-Lescure A, Hugh J, Loret C, Rupin M, Blitz S, Jacobs P, Murawsky M, Riva A, Vogel C; Breast Cancer International Research Group 001 Investigators. Adjuvant docetaxel for node-positive breast cancer. N Engl J Med. 2005 Jun 2;352(22):2302-13. doi: 10.1056/NEJMoa043681. PMID 15930421
- [Derived] Mackey JR, Martin M, Pienkowski T, Rolski J, Guastalla JP, Sami A, Glaspy J, Juhos E, Wardley A, Fornander T, Hainsworth J, Coleman R, Modiano MR, Vinholes J, Pinter T, Rodriguez-Lescure A, Colwell B, Whitlock P, Provencher L, Laing K, Walde D, Price C, Hugh JC, Childs BH, Bassi K, Lindsay MA, Wilson V, Rupin M, Houe V, Vogel C; TRIO/BCIRG 001 investigators. Adjuvant docetaxel, doxorubicin, and cyclophosphamide in node-positive breast cancer: 10-year follow-up of the phase 3 randomised BCIRG 001 trial. Lancet Oncol. 2013 Jan;14(1):72-80. doi: 10.1016/S1470-2045(12)70525-9. Epub 2012 Dec 12. PMID 23246022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 1997 and June 1999, 1491 women from 20 countries were enrolled in the study. The last patient last visit occurred in January 2010.
Pre-assignment Details: Eleven women (1 who had been randomly assigned to receive TAC and 10 assigned to receive FAC) did not receive any treatment for the following reasons: 8 withdrew consent, 1 was lost to follow-up, and 2 did not receive treatment for other reasons. In total 1480 patients (744 in the TAC group and 736 in the FAC group) were treated.
Groups:
- TAC (Docetaxel): docetaxel in combination with doxorubicin and cyclophosphamide
- FAC (5-fluorouracil): 5-fluorouracil in combination with doxorubicin and cyclophosphamide
Period: Overall Study
Arm/Group | TAC (Docetaxel) | FAC (5-fluorouracil)
Started | 745 | 746
Completed | 679 | 711
Not Completed | 66 | 35
Not completed — Adverse Event | 45 | 8
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Consent Withdrawn | 17 | 17
Not completed — Breast Cancer Relapse | 1 | 4
Not completed — Violation of Inclusion Criteria | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAC (Docetaxel) | FAC (5-fluorouracil) | Total
Number analyzed (Participants) | 745 | 746 | 1491
Age, Categorical [Count of Participants; unit: Participants]
  Between 18 and 65 years | 697 | 705 | 1402
  >=65 years | 48 | 41 | 89
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 745 | 746 | 1491
  Male | 0 | 0 | 0
Number of Positive Nodes [Number; unit: participants]
  1-3 Positive Nodes | 467 | 459 | 926
  4 or More Positive Nodes | 278 | 287 | 565

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Disease-Free Survival Events
Description: Disease-Free Survival (DFS)- are defined as local, regional or metastatic relapse or the date of second primary cancer or death from any cause whichever occurs first.
Time Frame: up to 10 year follow-up
Population: The study was originally designed to have 90% power to detect a 26% risk reduction of relapsing for TAC compared to FAC (hazard ratio=0.74)
Measure: Number; unit: Participants
Arm/Group | TAC (Docetaxel) | FAC (5-fluorouracil)
Number analyzed (Participants) | 745 | 746
Participants | 287 [0.579 to 0.650] | 333 [0.513 to 0.586]
Statistical Analysis 1: Comparison: TAC (Docetaxel) vs FAC (5-fluorouracil); Test type: Superiority or Other; p = 0.0043, Log Rank — Pairwise stratified log-rank test on the number of positive axillary nodes as per randomization; Cox Proportional Hazard = 0.795, 95% CI 2-sided [0.679 to 0.932]

2. Secondary Outcome: Number of Participants With Overall Survival Events
Description: Overall Survival - time from the date of randomization up to the date of death of any cause.
Time Frame: up to 10 year follow-up
Measure: Number; unit: Participants
Arm/Group | TAC (Docetaxel) | FAC (5-fluorouracil)
Number analyzed (Participants) | 745 | 746
Participants | 188 [0.724 to 0.786] | 241 [0.651 to 0.719]
Statistical Analysis 1: Comparison: TAC (Docetaxel) vs FAC (5-fluorouracil); Test type: Superiority or Other; p = 0.0020, Log Rank — Pairwise stratified log-rank test on the number of positive axillary nodes as per randomization; Cox Proportional Hazard = 0.742, 95% CI 2-sided [0.613 to 0.898]

3. Secondary Outcome: Number of Participants With Second Primary Malignancies (Toxicity)
Description: Toxicity (second primary malignancies)- defined as histopathologically proven cancer, excluding nonmelanomatous skin cancer, in situ carcinoma of the cervix, and in situ carcinoma of the breast.
Time Frame: up to 10 year follow-up
Measure: Number; unit: Participants
Arm/Group | TAC (Docetaxel) | FAC (5-fluorouracil)
Number analyzed (Participants) | 745 | 746
Participants | 67 | 66

ADVERSE EVENTS:
Time Frame: from date of randomization until the completion of the 10-year follow-up period.
Arm/Group | TAC (Docetaxel) | FAC (5-fluorouracil)
Serious Adverse Events (participants affected / at risk) | 267/744 | 67/736
Other Adverse Events (participants affected / at risk) | 744/744 | 734/736
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAC (Docetaxel) (N=744) | FAC (5-fluorouracil) (N=736)
Fever in absence of infection (General disorders) | 187 | 24
Pharyngitis (Infections and infestations) | 7 | 1
Pneumonia (Infections and infestations) | 4 | 2
Sepsis (Infections and infestations) | 4 | 2
Sinusitis (Infections and infestations) | 4 | 0
Urinary tract infection (Infections and infestations) | 4 | 3
Lung infection (Infections and infestations) | 3 | 0
Abscess (Infections and infestations) | 2 | 0
Catheter related infection (Infections and infestations) | 2 | 3
Catheter site cellulitis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 2 | 1
Lymphangitis (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0
Tonsillitis (Infections and infestations) | 2 | 0
Tooth abscess (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Abscess oral (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Candidiasis (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Oral infection (Infections and infestations) | 1 | 0
Pelvic inflammatory disease (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal skin infection (Infections and infestations) | 1 | 0
Trichomoniasis (Infections and infestations) | 1 | 0
Vulvitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Breast infection (Infections and infestations) | 0 | 1
Endometritis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Peritoneal infection (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 11 | 6
Nausea (Gastrointestinal disorders) | 8 | 3
Diarrhoea (Gastrointestinal disorders) | 6 | 1
Stomatitis (Gastrointestinal disorders) | 5 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Caecitis (Gastrointestinal disorders) | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer, obstructive (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Duodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Pyrexia (General disorders) | 6 | 2
Asthenia (General disorders) | 2 | 0
Chest pain (General disorders) | 2 | 0
Pain (General disorders) | 2 | 0
Injection site reaction (General disorders) | 1 | 0
Necrosis (General disorders) | 1 | 0
Catheter related complication (General disorders) | 0 | 1
Catheter site inflammation (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 1
Essential tremor (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 4 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 4
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 2
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 2 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Affective disorder (Psychiatric disorders) | 2 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Haemoglobin (Investigations) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAC (Docetaxel) (N=744) | FAC (5-fluorouracil) (N=736)
Any skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 734 | 718
Alopecia (Skin and subcutaneous tissue disorders) | 728 | 715
Skin disorder (Skin and subcutaneous tissue disorders) | 176 | 105
Nail disorder (Skin and subcutaneous tissue disorders) | 135 | 103
Any gastrointestinal disorders (Gastrointestinal disorders) | 713 | 709
Nausea (Gastrointestinal disorders) | 599 | 647
Stomatitis (Gastrointestinal disorders) | 508 | 374
Vomiting (Gastrointestinal disorders) | 327 | 436
Constipation (Gastrointestinal disorders) | 271 | 255
Diarrhoea (Gastrointestinal disorders) | 259 | 205
Dyspepsia (Gastrointestinal disorders) | 178 | 132
Haemorrhoids (Gastrointestinal disorders) | 57 | 35
Abdominal pain upper (Gastrointestinal disorders) | 44 | 22
Dry mouth (Gastrointestinal disorders) | 36 | 43
Any general disorders and administration site conditions (General disorders) | 673 | 610
Asthenia (General disorders) | 592 | 513
Pain (General disorders) | 312 | 264
Oedema peripheral (General disorders) | 250 | 91
Pyrexia (General disorders) | 152 | 87
Injection site reaction (General disorders) | 99 | 88
Chills (General disorders) | 53 | 29
Any nervous system disorders (Nervous system disorders) | 427 | 318
Dysgeusia (Nervous system disorders) | 206 | 112
Peripheral sensory neuropathy (Nervous system disorders) | 185 | 70
Headache (Nervous system disorders) | 153 | 169
Dizziness (Nervous system disorders) | 63 | 50
Any reproductive system and breast disorders (Reproductive system and breast disorders) | 307 | 268
Amenorrhoea (Reproductive system and breast disorders) | 212 | 136
Menstruation irregular (Reproductive system and breast disorders) | 211 | 165
Any infections and infestations (Infections and infestations) | 295 | 293
Nasopharyngitis (Infections and infestations) | 45 | 62
Upper respiratory tract infection (Infections and infestations) | 35 | 53
Any musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 290 | 152
Myalgia (Musculoskeletal and connective tissue disorders) | 199 | 73
Arthralgia (Musculoskeletal and connective tissue disorders) | 144 | 67
Any respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 280 | 196
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 117 | 64
Cough (Respiratory, thoracic and mediastinal disorders) | 100 | 72
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 60 | 53
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 39 | 27
Any vascular disorders (Vascular disorders) | 271 | 194
Hot flush (Vascular disorders) | 184 | 147
Flushing (Vascular disorders) | 49 | 26
Any psychiatric disorders (Psychiatric disorders) | 214 | 170
Insomnia (Psychiatric disorders) | 122 | 83
Affective disorder (Psychiatric disorders) | 82 | 76
Any eye disorders (Eye disorders) | 194 | 167
Lacrimation increased (Eye disorders) | 87 | 52
Any metabolism and nutrition disorders (Metabolism and nutrition disorders) | 185 | 140
Decreased appetite (Metabolism and nutrition disorders) | 161 | 130
Any investigations (Investigations) | 171 | 144
Weight increased (Investigations) | 131 | 108
Fever in absence of infection (General disorders) | 112 | 40
Any immune system disorders (Immune system disorders) | 93 | 24
Hypersensitivity (Immune system disorders) | 82 | 21
Any cardiac disorders (Cardiac disorders) | 77 | 51
Arrhythmia (Cardiac disorders) | 46 | 35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication of the study will be made without approval of the advisory board of the Breast Cancer International Research Group and Rhone- Poulenc Rorer.